CLINICAL TRIAL: NCT03150108
Title: A Phase 1, Open-label, Randomized, Cross-over Study to Evaluate the Pharmacokinetics, Safety, and Tolerability of a Single Dose of rhPTH(1-84) Administered Subcutaneously in Japanese Healthy Subjects Compared With Matched Non-Hispanic, Caucasian Healthy Adult Subjects and to Assess Dose Proportionality of 3 Doses of rhPTH(1-84) in the Japanese Subjects
Brief Title: Study of rhPTH(1-84) in Japanese Healthy Subjects Compared With Matched Caucasian Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SHP634-102
Record Dates: First submitted 2017-05-01; First posted 2017-05-12 (Actual); Results first posted 2019-07-12 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2021-05

CONDITIONS: Hypoparathyroidism
MeSH Terms: conditions — Hypoparathyroidism

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Non-Hispanic Caucasians (Experimental): Subjects will receive single dose of 100 microgram (mcg) rhPTH(1-84) subcutaneous (SC) injection on Day 1.
  Interventions: Drug: rhPTH(1-84)
- Participants of Japanese Descent (Experimental): Subjects will receive single dose of 100 mcg rhPTH(1-84) SC injection on Day 1; On days 4 and 7, either 25 mcg or 50 mcg SC injection. A washout period of 73 hours will be maintained between each single doses (100 mcg, 50 mcg and 25 mcg) in a cross-over fashion.
  Interventions: Drug: rhPTH(1-84)

INTERVENTIONS:
Drug: rhPTH(1-84) — 25 mcg rhPTH(1-84) SC injection
  Arms: Participants of Japanese Descent
Drug: rhPTH(1-84) — 50 mcg rhPTH(1-84) SC injection
  Arms: Participants of Japanese Descent
Drug: rhPTH(1-84) — 100 mcg rhPTH(1-84) SC injection
  Arms: Non-Hispanic Caucasians

SUMMARY:
The purpose of this study is to compare how rhPTH(1-84) affects the body between healthy adults of Japanese descent and matched, healthy Caucasian adults.

ELIGIBILITY:
Inclusion Criteria:

* Ability to voluntarily provide written, signed, and dated informed consent as applicable to participate in the study.
* An understanding, ability, and willingness to fully comply with study procedures and restrictions.
* Age 18-65 inclusive at the time of consent. The date of signature of the informed consent is defined as the beginning of the screening period. This inclusion criterion will only be assessed at the first screening visit.
* Subjects must be either:

  * A subject of Japanese descent born in Japan, who has resided outside of Japan for no longer than 5 years and is of Japanese parentage, defined as having 2 Japanese parents, and 4 Japanese grandparents, all born in Japan.
  * A non-hispanic, Caucasian subject who has 2 non-hispanic, Caucasian parents and 4 non-hispanic, Caucasian grandparents.
* Male or nonpregnant, nonlactating female who agrees to comply with any applicable contraceptive requirements of the protocol or females of nonchildbearing potential.
* Considered "healthy" by the investigator. Healthy status is defined by absence of evidence of any active or chronic disease following a detailed medical and surgical history, a complete physical examination including vital signs, 12-lead electrocardiogram (ECG), hematology, blood chemistry, and urinalysis.
* Body mass index between 18.5 and 28 kilogram per square meter (kg/m^2), inclusive, with a body weight greater than or equal to (>=) 45 kg (99 pounds [lbs]). This inclusion criterion will only be assessed at the first screening visit.
* Willing and able to consume standardized meals during the confinement period of the study. All subjects will be required to consume the identical meals on study days when serial pharmacokinetic (PK) and pharmacodynamic (PD) blood samples are collected.
* A clinical safety laboratory parameter of hemoglobin greater than (>) 11.7 gram per deciliter (g/dl) (females) or 13.1 g/dl (males) and less than (<) 16 g/dl (females) or 17.4 g/dl (males) or, if out of this range, deemed not clinically significant by the principal investigator.
* Total serum calcium within laboratory normal limits.
* Serum parathyroid hormone (PTH) levels within laboratory normal limits.

Exclusion Criteria:

* History of any hematological, hepatic, respiratory, cardiovascular, renal, neurological or psychiatric disease, gall bladder removal, or current or recurrent disease that could affect the action, absorption, or disposition of the investigational product, or clinical or laboratory assessments.
* Current or relevant history of physical or psychiatric illness, any medical disorder that may require treatment or make the subject unlikely to fully complete the study, or any condition that presents undue risk from the investigational product or procedures.
* Known or suspected intolerance or hypersensitivity to the investigational product(s), closely-related compounds, or any of the stated ingredients.
* Significant illness, as judged by the investigator, within 2 weeks of the first dose of investigational product.
* Known history of alcohol or other substance abuse within the last year.
* Donation of blood or blood products (Example (eg), plasma or platelets) within 60 days prior to receiving the first dose of investigational product.
* Use of the following prior to administration of investigational product within:

  * 30 days - loop diuretics, lithium, antacids, systemic corticosteroids (medical judgment is required by the investigator. Primarily high doses of systemic corticosteroids [eg, prednisone] should be excluded. Stable doses of hydrocortisone [eg, as treatment for Addison's disease] may be acceptable).
  * 3 months - calcitonin, cinacalcet hydrochloride, treatment with rhPTH(1-84) or N-terminal PTH or PTH-related peptide fragments or analogs.
  * For females: changes in hormone replacement therapy within 3 months are excluded. Stable (≥3 months) hormone replacement therapy is acceptable.
  * 6 months - fluoride tablets, oral bisphosphonates, methotrexate, growth hormone, digoxin, raloxifene or similar selective estrogen receptor modulators (SERMs).
  * 12 months - intravenous bisphosphonates, drug or alcohol abuse, as determined by the investigator.
* Confirmed systolic blood pressure (BP) >39 millimeter of mercury (mmHg) or <89 mmHg, and diastolic BP >89 mmHg or <49 mmHg.
* Twelve-lead ECG demonstrating measure of time between the start of the Q wave and the end of the T wave using Fridericia's formula in an electrocardiogram (QTcF) >450 milliseconds (msec) at screening. If QTcF exceeds 450 msec, the ECG should be repeated 2 more times and the average of the 3 QTcF values should be used to determine the subject's eligibility.
* Positive screen for drugs of abuse at screening or drugs of abuse or alcohol on Day -1.
* Male subjects who consume more than 21 units of alcohol per week or 3 units per day. Female subjects who consume more than 14 units of alcohol per week or 2 units per day. (1 alcohol unit=1 beer or 1 wine (5 ounce (oz) per 150 milliliter (mL)) or 1 liquor (1.5oz/40 mL) or 0.75 oz alcohol).
* Positive human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV) antibody screen.
* Use of tobacco in any form (eg, smoking or chewing) or other nicotine-containing products in any form (eg, gum, patch). Ex-users must report that they have stopped using tobacco for at least 30 days prior to receiving the first dose of investigational product.
* Routine consumption of more than 2 units of caffeine per day or subjects who experience caffeine withdrawal headaches. (1 caffeine unit is contained in the following items: one 6 oz (180 mL) cup of coffee, two 12 oz (360 mL) cans of cola, one 12 oz cup of tea, three 1 oz (85 g) chocolate bars. Decaffeinated coffee, tea, or cola are not considered to contain caffeine).
* Prior screen failure, randomization, participation, or enrollment in this study or prior exposure to any exogenous PTH, PTH fragments or analogs.
* Current use of any medication (including over-the-counter, herbal, or homeopathic preparations; with the exception of hormonal replacement therapy or hormonal contraceptives and occasional use of ibuprofen and acetaminophen). Current use is defined as use within 14 days of the first dose of investigational product.
* History of abnormalities of calcium homeostasis including hyperparathyroidism, hypoparathyroidism, hyperthyroidism, osteoporosis, Cushing's syndrome, hypercalcemia, hypocalcemia, or any other calcium disorder.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-05-16 (Actual); Primary Completion 2017-06-26 (Actual); Study Completion 2017-06-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Glendale Adventist Medical Center, Glendale, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at a single center in United States between 19 April 2017 (first participant first visit) and 26 Jun 2017 (last participant last visit).
Pre-assignment Details: A total of 24 participants (12 non-Hispanic healthy volunteer Caucasian participants and 12 healthy Japanese participants) were enrolled and randomized to study treatment.
Groups:
- Non-Hispanic Caucasians: Participants (who have 2 non-Hispanic Caucasian parents and 4 non-Hispanic Caucasian grandparents) matched to participants of Japanese descent based on sex (1:1 male: female), age (+/-7 years), and body mass index (+/-15%) received a single subcutaneous (SC) injection of 100 microgram (mcg) recombinant human parathyroid hormone (rhPTH[1-84]) on Day 1.
- Participants of Japanese Descent: Participants (born in Japan, who have resided outside of Japan for no longer than 5 years and were of Japanese parentage, defined as having 2 Japanese parents, and 4 Japanese grandparents, all born in Japan) received a single SC injection of 100 mcg rhPTH(1-84) on Day 1, then followed by either 25 mcg or 50 mcg SC injection on Days 4 and 7 in a cross-over fashion. A washout period of 73 hours was maintained between each single doses (100 mcg, 50 mcg and 25 mcg).
Period: Overall Study
Arm/Group | Non-Hispanic Caucasians | Participants of Japanese Descent
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety set included enrolled participants who received at least 1 dose of rhPTH(1-84).
Groups:
- Non-Hispanic Caucasians: Participants (who have 2 non-Hispanic Caucasian parents and 4 non-Hispanic Caucasian grandparents) matched to participants of Japanese descent based on sex (1:1 male: female), age (+/-7 years), and body mass index (+/-15%) received a single SC injection of 100 mcg rhPTH[1-84] on Day 1.
- Total: Total of all reporting groups
Arm/Group | Non-Hispanic Caucasians | Participants of Japanese Descent | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Continuous [Mean (Standard Deviation); unit: Years] | 40.3 (9.01) | 41.3 (10.40) | 40.8 (9.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 10 | 10 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 12 | 12 | 24
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 12 | 12
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 12 | 0 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Baseline-adjusted Cmax of PTH(1-84)
Description: Baseline-adjusted maximum observed drug concentration (Cmax) of PTH(1-84) in plasma was reported. The dispersion measure Geometric Coefficient of Variation was reported in percent (%).
Time Frame: 30 and 90 minutes (min) Pre-dose, 10, 20, 30, 45 min, 1, 1.25, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16 and 24 hours (h) Post-dose
Population: The pharmacokinetic (PK) set consisted of participants who received at least 1 dose of rhPTH(1-84) and had at least 1 evaluable post-dose PK concentration value.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Picogram per milliliter (pg/mL)
Groups:
- Non-Hispanic Caucasians: 100 mcg rhPTH(1-84): Participants (who have 2 non-Hispanic Caucasian parents and 4 non-Hispanic Caucasian grandparents) matched to participants of Japanese descent based on sex (1:1 male: female), age (+/-7 years), and body mass index (+/-15%) received a single subcutaneous (SC) injection of 100 microgram (mcg) recombinant human parathyroid hormone (rhPTH[1-84]) on Day 1.
- Participants of Japanese Descent: 100 mcg rhPTH(1-84): Participants (born in Japan, who have resided outside of Japan for no longer than 5 years and were of Japanese parentage, defined as having 2 Japanese parents, and 4 Japanese grandparents, all born in Japan) received a single SC injection of 100 mcg rhPTH(1-84) on Day 1.
- Participants of Japanese Descent: 50 mcg rhPTH(1-84): Participants (born in Japan, who have resided outside of Japan for no longer than 5 years and were of Japanese parentage, defined as having 2 Japanese parents, and 4 Japanese grandparents, all born in Japan) received a single SC injection of 50 mcg rhPTH(1-84) on Day 4 or 7.
- Participants of Japanese Descent: 25 mcg rhPTH(1-84): Participants (born in Japan, who have resided outside of Japan for no longer than 5 years and were of Japanese parentage, defined as having 2 Japanese parents, and 4 Japanese grandparents, all born in Japan) received a single SC injection of 25 mcg rhPTH(1-84) on Day 4 or 7.
Arm/Group | Non-Hispanic Caucasians: 100 mcg rhPTH(1-84) | Participants of Japanese Descent: 100 mcg rhPTH(1-84) | Participants of Japanese Descent: 50 mcg rhPTH(1-84) | Participants of Japanese Descent: 25 mcg rhPTH(1-84)
Number analyzed (Participants) | 12 | 12 | 12 | 12
Picogram per milliliter (pg/mL) | 295.662 (41.66) | 330.820 (29.44) | 175.468 (35.29) | 99.708 (22.02)
Statistical Analysis 1: Comparison: Non-Hispanic Caucasians: 100 mcg rhPTH(1-84) vs Participants of Japanese Descent: 100 mcg rhPTH(1-84); Test type: Equivalence — Welch's t-test with Satterthwaite's approximation to the degrees of freedom was used to compare the log transformed Cmax values of both ethnic groups at 100 mcg dose and the results were back-transformed to get the estimates for the geometric means and for the ratio of geometric means (Japanese/Caucasian), and 90% confidence interval (CI); Geometric mean ratio = 1.119, 90% CI 2-sided [0.875 to 1.430]
Statistical Analysis 2: Comparison: Participants of Japanese Descent: 100 mcg rhPTH(1-84) vs Participants of Japanese Descent: 50 mcg rhPTH(1-84) vs Participants of Japanese Descent: 25 mcg rhPTH(1-84); Dose proportionality was assessed for baseline-adjusted Cmax using the power model. The power model assumes a linear relationship between the natural log transformed parameter and the natural log transformed dose. The fold increase in PK parameters with doubling the dose and the 90% CIs were calculated; Test type: Other — Dose proportionality; Increase in Cmax per Dose Doubling = 1.76, 90% CI 2-sided [1.52 to 2.03] — Linear model of log transformed PK parameters at all doses in Japanese descent, including log transformed dose, period, sequence as fixed effects, and intercept as a random effect accounting for each participant within sequence as their own control

2. Primary Outcome: Baseline-adjusted Tmax of PTH(1-84)
Description: Baseline-adjusted time to reach maximum observed drug concentration (Tmax) of PTH(1-84) in plasma was reported.
Time Frame: 30 and 90 min Pre-dose,10, 20, 30, 45 min, 1, 1.25, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16 and 24 h Post-dose
Population: The PK set consisted of participants who received at least 1 dose of rhPTH(1-84) and had at least 1 evaluable post-dose PK concentration value.
Measure: Median (Full Range); unit: Hour (h)
Arm/Group | Non-Hispanic Caucasians: 100 mcg rhPTH(1-84) | Participants of Japanese Descent: 100 mcg rhPTH(1-84) | Participants of Japanese Descent: 50 mcg rhPTH(1-84) | Participants of Japanese Descent: 25 mcg rhPTH(1-84)
Number analyzed (Participants) | 12 | 12 | 12 | 12
Hour (h) | 0.415 [0.17 to 3.00] | 1.000 [0.17 to 4.00] | 1.385 [0.50 to 2.50] | 1.240 [0.17 to 2.00]

3. Primary Outcome: Baseline-adjusted AUC(Last) of PTH(1-84) in Plasma
Description: Baseline-adjusted area under the curve from the time of dosing to the last measurable concentration (AUC(last)) of PTH(1-84) was reported. The dispersion measure Geometric Coefficient of Variation was reported in percent (%).
Time Frame: 30 and 90 min Pre-dose,10, 20, 30, 45 min, 1, 1.25, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16 and 24 h Post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*picogram per milliliter (h*pg/mL)
Arm/Group | Non-Hispanic Caucasians: 100 mcg rhPTH(1-84) | Participants of Japanese Descent: 100 mcg rhPTH(1-84) | Participants of Japanese Descent: 50 mcg rhPTH(1-84) | Participants of Japanese Descent: 25 mcg rhPTH(1-84)
Number analyzed (Participants) | 12 | 12 | 12 | 12
Hour*picogram per milliliter (h*pg/mL) | 1037.63 (31.0) | 1027.81 (32.6) | 602.06 (30.6) | 255.67 (28.7)
Statistical Analysis 1: Comparison: Non-Hispanic Caucasians: 100 mcg rhPTH(1-84) vs Participants of Japanese Descent: 100 mcg rhPTH(1-84); Test type: Equivalence — Welch's t-test with Satterthwaite's approximation to the degrees of freedom was used to compare the log transformed AUClast values of both ethnic groups at 100 mcg dose and the results were back-transformed to get the estimates for the geometric means and for the ratio of geometric means (Japanese/Caucasian), and 90% CI; Geometric mean ratio = 0.99, 90% CI 2-sided [0.80 to 1.23]
Statistical Analysis 2: Comparison: Participants of Japanese Descent: 100 mcg rhPTH(1-84) vs Participants of Japanese Descent: 50 mcg rhPTH(1-84) vs Participants of Japanese Descent: 25 mcg rhPTH(1-84); Dose proportionality was assessed for baseline-adjusted AUClast using the power model. The power model assumes a linear relationship between the natural log transformed parameter and the natural log transformed dose. The fold increase in PK parameters with doubling the dose and the 90% CIs were calculated; Test type: Other — Dose proportionality; Increase in AUClast per Dose Doubling = 2.35, 90% CI [2.06 to 2.70] — [estimate comment as in outcome 1, analysis 2]

4. Primary Outcome: Baseline-adjusted AUC(0-8) of PTH(1-84) in Plasma
Description: Baseline-adjusted area under the concentration versus time curve from the time of dosing to 8 hours post dose (AUC(0-8)) of PTH(1-84) was reported. The dispersion measure Geometric Coefficient of Variation was reported in percent (%).
Time Frame: 30 and 90 min Pre-dose,10, 20, 30, 45 min, 1, 1.25, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16 and 24 h Post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*pg/mL
Groups:
- Non-Hispanic Caucasians:100 mcg rhPTH(1-84): Participants (who have 2 non-Hispanic Caucasian parents and 4 non-Hispanic Caucasian grandparents) matched to participants of Japanese descent based on sex (1:1 male: female), age (+/-7 years), and body mass index (+/-15%) received a single subcutaneous (SC) injection of 100 microgram (mcg) recombinant human parathyroid hormone (rhPTH[1-84]) on Day 1.
Arm/Group | Non-Hispanic Caucasians:100 mcg rhPTH(1-84) | Participants of Japanese Descent: 100 mcg rhPTH(1-84) | Participants of Japanese Descent: 50 mcg rhPTH(1-84) | Participants of Japanese Descent: 25 mcg rhPTH(1-84)
Number analyzed (Participants) | 12 | 12 | 12 | 12
h*pg/mL | 956.63 (32.8) | 1033.62 (31.4) | 554.23 (30.8) | 248.38 (19.7)
Statistical Analysis 1: Comparison: Non-Hispanic Caucasians:100 mcg rhPTH(1-84) vs Participants of Japanese Descent: 100 mcg rhPTH(1-84); Test type: Equivalence — Welch's t-test with Satterthwaite's approximation to the degrees of freedom was used to compare the log transformed AUC0-8 values of both ethnic groups at 100 mcg dose and the results were back-transformed to get the estimates for the geometric means and for the ratio of geometric means (Japanese/Caucasian), and 90% CI; Geometric mean ratio = 1.08, 90% CI 2-sided [0.87 to 1.35]
Statistical Analysis 2: Comparison: Participants of Japanese Descent: 100 mcg rhPTH(1-84) vs Participants of Japanese Descent: 50 mcg rhPTH(1-84) vs Participants of Japanese Descent: 25 mcg rhPTH(1-84); Dose proportionality was assessed for baseline-adjusted AUC0-8 using the power model. The power model assumes a linear relationship between the natural log transformed parameter and the natural log transformed dose. The fold increase in PK parameters with doubling the dose and the 90% CIs were calculated; Test type: Other — Dose proportionality; Increase in AUC0-8 per Dose Doubling = 2.23, 90% CI 2-sided [1.98 to 2.51] — [estimate comment as in outcome 1, analysis 2]

5. Primary Outcome: Baseline-adjusted AUC(0-inf) of PTH(1-84) in Plasma
Description: Baseline-adjusted area under the concentration versus time curve extrapolated to infinity (AUC(0-inf)) of PTH(1-84) was reported. The dispersion measure Geometric Coefficient of Variation was reported in percent (%).
Time Frame: 30 and 90 min Pre-dose,10, 20, 30, 45 min, 1, 1.25, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16 and 24 h Post-dose
Population: The PK set consisted of participants who received at least 1 dose of rhPTH(1-84) and had at least 1 evaluable post-dose PK concentration value. Here number of participants analyzed indicates the participants evaluable for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*pg/mL
Arm/Group | Non-Hispanic Caucasians: 100 mcg rhPTH(1-84) | Participants of Japanese Descent: 100 mcg rhPTH(1-84) | Participants of Japanese Descent: 50 mcg rhPTH(1-84) | Participants of Japanese Descent: 25 mcg rhPTH(1-84)
Number analyzed (Participants) | 8 | 10 | 9 | 10
h*pg/mL | 1028.29 (37.0) | 1039.34 (29.8) | 589.25 (31.6) | 249.51 (21.9)
Statistical Analysis 1: Comparison: Non-Hispanic Caucasians: 100 mcg rhPTH(1-84) vs Participants of Japanese Descent: 100 mcg rhPTH(1-84); Test type: Equivalence — Welch's t-test with Satterthwaite's approximation to the degrees of freedom was used to compare the log transformed AUC0-inf values of both ethnic groups at 100 mcg dose and the results were back-transformed to get the estimates for the geometric means and for the ratio of geometric means (Japanese/Caucasian), and 90% CI; Geometric mean ratio = 1.01, 90% CI 2-sided [0.77 to 1.33]
Statistical Analysis 2: Comparison: Participants of Japanese Descent: 100 mcg rhPTH(1-84) vs Participants of Japanese Descent: 50 mcg rhPTH(1-84) vs Participants of Japanese Descent: 25 mcg rhPTH(1-84); Dose proportionality was assessed for baseline-adjusted AUC0-inf using the power model. The power model assumes a linear relationship between the natural log transformed parameter and the natural log transformed dose. The fold increase in PK parameters with doubling the dose and the 90% CIs were calculated; Test type: Other — Dose proportionality; Increase in AUC0-inf per Dose Doubling = 2.31, 90% CI 2-sided [1.96 to 2.71] — [estimate comment as in outcome 1, analysis 2]

6. Primary Outcome: Baseline- Adjusted % of AUC(0-Inf) Extra of PTH(1-84) in Plasma
Description: Baseline-adjusted % of AUC extrapolated from the last measurable concentration to infinity over (AUC(0-Inf)) of PTH(1-84) in plasma was reported. The dispersion measure Geometric Coefficient of Variation was reported in percent (%).
Time Frame: 30 and 90 min Pre-dose,10, 20, 30, 45 min, 1, 1.25, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16 and 24 h Post-dose
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage of AUC
Arm/Group | Non-Hispanic Caucasians:100 mcg rhPTH(1-84) | Participants of Japanese Descent: 100 mcg rhPTH(1-84) | Participants of Japanese Descent: 50 mcg rhPTH(1-84) | Participants of Japanese Descent: 25 mcg rhPTH(1-84)
Number analyzed (Participants) | 8 | 10 | 9 | 10
Percentage of AUC | 1.416 (198.59) | 0.932 (330.55) | 1.555 (173.86) | 3.015 (135.99)

7. Primary Outcome: Baseline-adjusted Lambda_z of PTH(1-84) in Plasma
Description: Baseline-adjusted Lambda z associated with the terminal (log-linear) portion of the curve for PTH(1-84) in plasma was reported. The dispersion measure Geometric Coefficient of Variation was reported in percent (%).
Time Frame: 30 and 90 min Pre-dose,10, 20, 30, 45 min, 1, 1.25, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16 and 24 h Post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Per hour (1/h)
Arm/Group | Non-Hispanic Caucasians:100 mcg rhPTH(1-84) | Participants of Japanese Descent: 100 mcg rhPTH(1-84) | Participants of Japanese Descent: 50 mcg rhPTH(1-84) | Participants of Japanese Descent: 25 mcg rhPTH(1-84)
Number analyzed (Participants) | 8 | 10 | 9 | 10
Per hour (1/h) | 0.4496 (67.730) | 0.6672 (35.835) | 0.5714 (65.437) | 0.8277 (57.118)

8. Primary Outcome: Baseline-adjusted t1/2 of PTH(1-84) in Plasma
Description: Baseline-adjusted Terminal Half-life (t1/2) of PTH(1-84) in plasma was reported.
Time Frame: 30 and 90 min Pre-dose,10, 20, 30, 45 min, 1, 1.25, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16 and 24 h Post-dose
Population: as for outcome 5
Measure: Median (Full Range); unit: Hour (h)
Arm/Group | Non-Hispanic Caucasians:100 mcg rhPTH(1-84) | Participants of Japanese Descent: 100 mcg rhPTH(1-84) | Participants of Japanese Descent: 50 mcg rhPTH(1-84) | Participants of Japanese Descent: 25 mcg rhPTH(1-84)
Number analyzed (Participants) | 8 | 10 | 9 | 10
Hour (h) | 1.390 [0.68 to 4.74] | 1.060 [0.65 to 1.71] | 1.020 [0.69 to 3.57] | 0.950 [0.30 to 1.88]

9. Primary Outcome: Baseline-adjusted CL/F of PTH(1-84) in Plasma
Description: Baseline-adjusted apparent clearance (CL/F) of PTH(1-84) in plasma was reported. The dispersion measure Geometric Coefficient of Variation was reported in percent (%).
Time Frame: 30 and 90 min Pre-dose,10, 20, 30, 45 min, 1, 1.25, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16 and 24 h Post-dose
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter per hour (L/h)
Arm/Group | Non-Hispanic Caucasians:100 mcg rhPTH(1-84) | Participants of Japanese Descent: 100 mcg rhPTH(1-84) | Participants of Japanese Descent: 50 mcg rhPTH(1-84) | Participants of Japanese Descent: 25 mcg rhPTH(1-84)
Number analyzed (Participants) | 8 | 10 | 9 | 10
Liter per hour (L/h) | 97.25 (37.0) | 96.22 (29.8) | 84.84 (31.6) | 100.18 (21.9)

10. Primary Outcome: Baseline-adjusted Vdz/F of PTH(1-84) in Plasma
Description: Baseline-adjusted apparent volume of distribution (Vdz/F) of PTH(1-84) in plasma was reported. The dispersion measure Geometric Coefficient of Variation was reported in percent (%).
Time Frame: 30 and 90 min Pre-dose,10, 20, 30, 45 min, 1, 1.25, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16 and 24 h Post-dose
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters (L)
Arm/Group | Non-Hispanic Caucasians:100 mcg rhPTH(1-84) | Participants of Japanese Descent: 100 mcg rhPTH(1-84) | Participants of Japanese Descent: 50 mcg rhPTH(1-84) | Participants of Japanese Descent: 25 mcg rhPTH(1-84)
Number analyzed (Participants) | 8 | 10 | 9 | 10
Liters (L) | 216.30 (93.9) | 144.18 (54.7) | 148.50 (71.9) | 121.02 (57.7)

11. Secondary Outcome: Original Cmax of PTH(1-84) in Plasma
Description: Original maximum observed drug concentration (Cmax) of PTH(1-84) in plasma was reported. The dispersion measure Geometric Coefficient of Variation was reported in percent (%).
Time Frame: 30 and 90 min Pre-dose,10, 20, 30, 45 min, 1, 1.25, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16 and 24 h Post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | Non-Hispanic Caucasians:100 mcg rhPTH(1-84) | Participants of Japanese Descent: 100 mcg rhPTH(1-84) | Participants of Japanese Descent: 50 mcg rhPTH(1-84) | Participants of Japanese Descent: 25 mcg rhPTH(1-84)
Number analyzed (Participants) | 12 | 12 | 12 | 12
pg/mL | 324.43 (36.2) | 365.52 (27.3) | 206.05 (29.6) | 129.74 (21.1)
Statistical Analysis 1: Comparison: Non-Hispanic Caucasians:100 mcg rhPTH(1-84) vs Participants of Japanese Descent: 100 mcg rhPTH(1-84); Test type: Equivalence — Welch's t-test with Satterthwaite's approximation to the degrees of freedom was used to compare the log transformed Cmax values of both ethnic groups at 100 mcg dose and the results were back-transformed to get the estimates for the geometric means and for the ratio of geometric means (Japanese/Caucasian), and 90% CI; Geometric Mean Ratio = 1.13, 90% CI 2-sided [0.90 to 1.40]

12. Secondary Outcome: Original Tmax of PTH(1-84)
Description: The original time to reach maximum observed drug concentration (Tmax) of PTH(1-84) in plasma was reported.
Time Frame: 30 and 90 min Pre-dose,10, 20, 30, 45 min, 1, 1.25, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16 and 24 h Post-dose
Population: as for outcome 2
Measure: Median (Full Range); unit: Hour (h)
Arm/Group | Non-Hispanic Caucasians:100 mcg rhPTH(1-84) | Participants of Japanese Descent: 100 mcg rhPTH(1-84) | Participants of Japanese Descent: 50 mcg rhPTH(1-84) | Participants of Japanese Descent: 25 mcg rhPTH(1-84)
Number analyzed (Participants) | 12 | 12 | 12 | 12
Hour (h) | 0.415 [0.17 to 3.00] | 1.000 [0.17 to 4.00] | 1.385 [0.50 to 2.50] | 1.240 [0.17 to 2.00]

13. Secondary Outcome: Original AUClast of PTH(1-84) in Plasma
Description: Original area under the curve from the time of dosing to the last measurable concentration (AUClast) of PTH(1-84) was reported. The dispersion measure Geometric Coefficient of Variation was reported in percent (%).
Time Frame: 30 and 90 min Pre-dose,10, 20, 30, 45 min, 1, 1.25, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16 and 24 h Post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*pg/mL
Arm/Group | Non-Hispanic Caucasians:100 mcg rhPTH(1-84) | Participants of Japanese Descent: 100 mcg rhPTH(1-84) | Participants of Japanese Descent: 50 mcg rhPTH(1-84) | Participants of Japanese Descent: 25 mcg rhPTH(1-84)
Number analyzed (Participants) | 12 | 12 | 12 | 12
h*pg/mL | 1685.62 (18.2) | 1823.70 (23.7) | 1300.09 (21.7) | 959.49 (26.1)
Statistical Analysis 1: Comparison: Non-Hispanic Caucasians:100 mcg rhPTH(1-84) vs Participants of Japanese Descent: 100 mcg rhPTH(1-84); Test type: Equivalence — [test comment as in outcome 11, analysis 1]; Geometric Mean Ratio = 1.08, 90% CI 2-sided [0.93 to 1.25]

14. Secondary Outcome: AUClast of Albumin-corrected Calcium, Serum Total Calcium and Phosphate Levels After Intake of PTH(1-84)
Description: Area under the curve from the time of dosing to the last measurable concentration of albumin-corrected calcium, serum total calcium and phosphate levels after intake of PTH(1-84) was reported. The dispersion measure Geometric Coefficient of Variation was reported in percent (%).
Time Frame: Non-Hispanic Caucasians: 30 mins predose, 4, 8 and 12 h (Day 1),24 h (Day 2) Japanese Descents: 30 mins predose, 4, 8 and 12 h (Days 1, 4, 7), 24 h (Days 2, 5, 8)
Population: The pharmacodynamic (PD) set consisted of participants who received at least 1 dose of rhPTH(1-84) and had at least 1 evaluable post-dose PD concentration value.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours * millimoles per liter (h×mmol/L)
Groups:
- Non-Hispanic Caucasians:100 mcg rhPTH(1-84); Participants of Japanese Descent: 100 mcg rhPTH(1-84): Participants received a single SC injection of 100 mcg rhPTH(1-84) on Day 1.
- Participants of Japanese Descent: 50 mcg rhPTH(1-84): Participants received a single SC injection of 50 mcg rhPTH(1-84) on Day 4 or 7.
- Participants of Japanese Descent: 25 mcg rhPTH(1-84): Participants received a single SC injection of 25 mcg rhPTH(1-84) on Day 4 or 7.
Arm/Group | Non-Hispanic Caucasians:100 mcg rhPTH(1-84) | Participants of Japanese Descent: 100 mcg rhPTH(1-84) | Participants of Japanese Descent: 50 mcg rhPTH(1-84) | Participants of Japanese Descent: 25 mcg rhPTH(1-84)
Number analyzed (Participants) | 12 | 12 | 12 | 12
Hours * millimoles per liter (h×mmol/L)
  Albumin-corrected Calcium | 52.94 (2.5) | 53.22 (2.3) | 52.94 (2.5) | 52.61 (3.1)
  Serum Total Calcium | 54.21 (2.7) | 54.62 (1.5) | 54.12 (2.6) | 53.62 (3.5)
  Serum Phosphate | 27.21 (10.5) | 28.85 (10.2) | 28.60 (7.8) | 29.57 (7.6)

15. Secondary Outcome: TEmax After Intake of PTH(1-84) on Albumin-corrected Calcium, Serum Total Calcium and Serum Phosphate Levels
Description: The time to maximum effect (TEmax) of PTH(1-84) on albumin-corrected calcium, serum total calcium and serum phosphate levels were reported.
Time Frame: as for outcome 14
Population: The PD set consisted of participants who received at least 1 dose of rhPTH(1-84) and had at least 1 evaluable post-dose PD concentration value.
Measure: Median (Full Range); unit: Hour (h)
Arm/Group | Non-Hispanic Caucasians:100 mcg rhPTH(1-84) | Participants of Japanese Descent: 100 mcg rhPTH(1-84) | Participants of Japanese Descent: 50 mcg rhPTH(1-84) | Participants of Japanese Descent: 25 mcg rhPTH(1-84)
Number analyzed (Participants) | 12 | 12 | 12 | 12
Hour (h)
  Albumin-corrected Calcium | 8.000 [4.00 to 12.02] | 8.000 [4.00 to 12.00] | 4.000 [0.00 to 8.00] | 4.000 [0.00 to 8.00]
  Serum Total Calcium | 8.000 [0.00 to 12.02] | 8.000 [4.00 to 12.00] | 8.000 [4.00 to 8.00] | 4.000 [0.00 to 12.02]
  Serum Phosphate | 8.010 [0.00 to 12.05] | 8.000 [4.00 to 11.98] | 8.000 [7.97 to 12.08] | 8.000 [0.00 to 12.02]

16. Secondary Outcome: Emax of PTH(1-84) on Albumin-corrected Calcium, Serum Total Calcium and Serum Phosphate Levels
Description: The maximum effect (Emax) of PTH(1-84) on albumin-corrected calcium, serum total calcium and serum phosphate levels were reported. The dispersion measure Geometric Coefficient of Variation was reported in percent (%).
Time Frame: as for outcome 14
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: millimoles per liter (mmol/L)
Arm/Group | Non-Hispanic Caucasians:100 mcg rhPTH(1-84) | Participants of Japanese Descent: 100 mcg rhPTH(1-84) | Participants of Japanese Descent: 50 mcg rhPTH(1-84) | Participants of Japanese Descent: 25 mcg rhPTH(1-84)
Number analyzed (Participants) | 12 | 12 | 12 | 12
millimoles per liter (mmol/L)
  Albumin-corrected Calcium | 2.287 (2.31) | 2.284 (2.46) | 2.283 (3.09) | 2.282 (2.34)
  Serum Total Calcium | 2.359 (3.49) | 2.347 (1.83) | 2.330 (2.60) | 2.322 (2.02)
  Serum Phosphate | 1.286 (11.88) | 1.325 (11.47) | 1.325 (7.94) | 1.383 (8.06)

17. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was defined as any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product and that did not necessarily have a causal relationship with this treatment.
Time Frame: From start of study drug administration to follow-up (up to 40 days)
Population: The safety set included enrolled participants who received at least 1 dose of rhPTH(1-84).
Measure: Count of Participants; unit: Participants
Arm/Group | Non-Hispanic Caucasians:100 mcg rhPTH(1-84) | Participants of Japanese Descent: 100 mcg rhPTH(1-84) | Participants of Japanese Descent: 50 mcg rhPTH(1-84) | Participants of Japanese Descent: 25 mcg rhPTH(1-84)
Number analyzed (Participants) | 12 | 12 | 12 | 12
Participants | 4 | 6 | 1 | 3

18. Secondary Outcome: Number of Participants With Clinically Significant Changes in Clinical Laboratory Tests Reported as Treatment-emergent Adverse Events (TEAEs)
Description: Clinical laboratory tests included hematology, chemistry, and urinalysis. Number of participants with clinically significant changes in clinical laboratory tests reported as TEAEs were reported.
Time Frame: Non-Hispanic Caucasians: 30 min pre-dose,24 h,32 days post-dose Japanese Descents: 30 min pre-dose,24 h post-dose on Days 1,4,7 and 32 days after last dose
Population: The safety set included enrolled participants who received at least 1 dose of rhPTH(1-84).
Measure: Count of Participants; unit: Participants
Arm/Group | Non-Hispanic Caucasians:100 mcg rhPTH(1-84) | Participants of Japanese Descent: 100 mcg rhPTH(1-84) | Participants of Japanese Descent: 50 mcg rhPTH(1-84) | Participants of Japanese Descent: 25 mcg rhPTH(1-84)
Number analyzed (Participants) | 12 | 12 | 12 | 12
Participants | 0 | 0 | 0 | 0

19. Secondary Outcome: Number of Participants With Clinically Significant Changes in Vital Signs Reported as Treatment-emergent Adverse Events (TEAEs)
Description: Vital signs were obtained while participant was supine. Vital signs included hematology, chemistry, and urinalysis. Number of participants with clinically significant changes in vital signs reported as TEAEs were reported.
Time Frame: Non-Hispanic Caucasians: 30 min pre-dose,1,4,8,24 h,32 days post-dose Japanese Descents: 30 min pre-dose,1,4,8,24 h post-dose on Days 1,4,7 and 32 days after last dose
Population: The safety set included enrolled participants who received at least 1 dose of rhPTH(1-84).
Measure: Count of Participants; unit: Participants
Arm/Group | Non-Hispanic Caucasians:100 mcg rhPTH(1-84) | Participants of Japanese Descent: 100 mcg rhPTH(1-84) | Participants of Japanese Descent: 50 mcg rhPTH(1-84) | Participants of Japanese Descent: 25 mcg rhPTH(1-84)
Number analyzed (Participants) | 12 | 12 | 12 | 12
Participants | 0 | 0 | 0 | 0

20. Secondary Outcome: Number of Participants With Clinically Significant Changes in Electrocardiogram (ECG) Results Reported as Treatment-emergent Adverse Events (TEAEs)
Description: Twelve-lead ECGs were performed in triplicate at each time point. For numeric ECG variables, the mean of the valid values at each time point was taken. Number of participants with clinically significant changes in ECGs reported as TEAEs were reported.
Time Frame: as for outcome 18
Population: The safety set included enrolled participants who received at least 1 dose of rhPTH(1-84).
Measure: Count of Participants; unit: Participants
Arm/Group | Non-Hispanic Caucasians:100 mcg rhPTH(1-84) | Participants of Japanese Descent: 100 mcg rhPTH(1-84) | Participants of Japanese Descent: 50 mcg rhPTH(1-84) | Participants of Japanese Descent: 25 mcg rhPTH(1-84)
Number analyzed (Participants) | 12 | 12 | 12 | 12
Participants | 0 | 0 | 0 | 0

21. Secondary Outcome: Number of Participants Who Reported Positive to Anti-Parathyroid Hormone Antibodies
Description: Number of participants who reported positive to anti-parathyroid hormone antibodies were reported.
Time Frame: Non-Hispanic Caucasians: 30 min pre-dose,32 days post-dose Japanese Descents: 30 min pre-dose on Days 1,4,7 and 32 days after last dose
Population: The safety set included enrolled participants who received at least 1 dose of rhPTH(1-84).
Measure: Count of Participants; unit: Participants
Arm/Group | Non-Hispanic Caucasians:100 mcg rhPTH(1-84) | Participants of Japanese Descent: 100 mcg rhPTH(1-84) | Participants of Japanese Descent: 50 mcg rhPTH(1-84) | Participants of Japanese Descent: 25 mcg rhPTH(1-84)
Number analyzed (Participants) | 12 | 12 | 12 | 12
Participants | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From start of study drug administration to follow-up (up to 40 days)
Groups:
- Non-Hispanic Caucasians:100 mcg rhPTH(1- 84); Participants of Japanese Descent: 100 mcg rhPTH(1-84): Participants received a single SC injection of 100 mcg rhPTH(1-84) on Day 1.
Arm/Group | Non-Hispanic Caucasians:100 mcg rhPTH(1- 84) | Participants of Japanese Descent: 100 mcg rhPTH(1-84) | Participants of Japanese Descent: 50 mcg rhPTH(1-84) | Participants of Japanese Descent: 25 mcg rhPTH(1-84)
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 4/12 | 6/12 | 1/12 | 3/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Non-Hispanic Caucasians:100 mcg rhPTH(1- 84) (N=12) | Participants of Japanese Descent: 100 mcg rhPTH(1-84) (N=12) | Participants of Japanese Descent: 50 mcg rhPTH(1-84) (N=12) | Participants of Japanese Descent: 25 mcg rhPTH(1-84) (N=12)
Nausea (Gastrointestinal disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sunburn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 3 (3) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.

DOCUMENTS (3):
  • Study Protocol: Original (2017-01-29): https://cdn.clinicaltrials.gov/large-docs/08/NCT03150108/Prot_000.pdf
  • Study Protocol: Amendment 1 (2017-03-21): https://cdn.clinicaltrials.gov/large-docs/08/NCT03150108/Prot_001.pdf
  • Statistical Analysis Plan (2017-06-12): https://cdn.clinicaltrials.gov/large-docs/08/NCT03150108/SAP_002.pdf